CLINICAL TRIAL: NCT01948661
Title: Randomized Window of Opportunity Trial of Anthocyanin Extract and Phospholipid Curcumin in Subjects With Colorectal Adenoma
Brief Title: Anthocyanin Extract and Phospholipid Curcumin in Colorectal Adenoma
Acronym: MIRACOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ente Ospedaliero Ospedali Galliera (Other)
Collaborators: Fondazione Umberto Veronesi (Other); Indena S.p.A (Industry)
Responsible Party: Principal Investigator, Andrea DeCensi, Medical Oncology Director, Ente Ospedaliero Ospedali Galliera
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GAL 02
Record Dates: First submitted 2013-01-18; First posted 2013-09-23 (Estimated); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Adenoma; Risk Reduction
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anthocyanins+Phospholipidic Curcumin (Experimental): Mirtoselect ® 500 mg tablet, 1000 mg (two oral tablets) per day and Meriva ®, 500 mg tablet, 1000 mg (two oral tablets) per day for 28 days
  Interventions: Dietary Supplement: Mirtoselect® + Meriva®
- placeboA + placeboB (Placebo Comparator): placeboA + placeboB per day for four weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Mirtoselect® + Meriva®
  Arms: Anthocyanins+Phospholipidic Curcumin
Dietary Supplement: Placebo
  Arms: placeboA + placeboB

SUMMARY:
It has been shown that curcumin and cyanidin-3-glucoside (C3G) have anticancer effects. In this clinical trial we compare the affect of their combination vs placebo in a four weeks intervention before endoscopic polypectomy.

DETAILED DESCRIPTION:
Colonic adenomatous polyps are pre cancer lesions and are used as intermediate markers for testing agents with potential cancer prevention.

Meriva© is a bioavailable form of curcumin, a polyphenolic compound obtained from turmeric (Curcuma longa L.) endowed with anti-inflammatory, antioxidant and antitumor effects. In vivo data indicate that curcumin formulated with phosphatidylcholine furnishes higher blood levels of parent agent than natural curcumin.

Mirtoselect©, an anthocyanin mixture from bilberry containing isolated cyanidin-3-glucoside (C3G), the most abundant anthocyanin in diet, prevents intestinal adenoma formation in the Apc(Min) mouse model.

The investigators hypothesize that the combination of both agents will decrease the expression of proteins involved in colon tumorigenesis relative to placebo.

The change of biomarker expression between pre-treatment biopsy and post-treatment endoscopic resection in the target adenoma and the normal rectal mucosa will be the response measures.

The primary response measure is the change of immunohistochemical (IHC) expression of β-catenin in adenomatous tissue and normal rectal mucosa. Secondary response measures are the changes of IHC Nuclear Factor-Kβ (NFKβ), cell proliferation by Ki-67 Labeling Index and apoptosis by P53 in adenomatous and adjacent normal mucosa.

The study design is a phase II, randomized, double blind, placebo controlled, window of opportunity trial of the combination of Mirtoselect 1 gr/day+Meriva 1 gr/day or placebo. Subjects with histological confirmation of colorectal adenomatous polyps >1 cm not suitable to immediate complete removal will be enrolled in a 4-week intervention trial before endoscopic polypectomy.

The demonstration of a biological activity of the two agent combination may provide the rationale for a phase III trial aimed at reducing the risk of colon cancer in high risk subjects.

ELIGIBILITY:
Inclusion criteria:

* Subjects with colorectal adenomatous polyps greater than 1 cm in maximum diameter not suitable to immediate complete removal;
* Normal renal and hepatic function;
* WHO Performance status=0;

Exclusion Criteria:

* Presence of hyperplastic polyps and/or flat adenomas;
* Subjects with pre-existing colorectal cancer;
* Presence of carcinomatous tissue in adenoma;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2022-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea DeCensi, MD, Principal Investigator — Medical Oncology Ente Ospedaliero Ospedali Galliera
Locations (4):
- Italy (4):
  - "Gastroenterologia d'urgenza ed Endoscopia digestiva" Ospedale di Lavagna ASL 4 Chiavarese, Chiavari
  - S.S. Gastroenterologia Ospedale Villa Scassi, ASL3 Genovese, Genoa
  - Medical Oncology Ente Ospedaliero Ospedali Galliera, Genova
  - Divisione di Prevenzione e Genetica Oncologica, IEO, Milan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 53 participants were contacted:
  * 8 refused to participate,
  * 45 signed the Informed Consent: 10 were not eligible and 35 were randomized
Groups:
- Experimental: Anthocyanins+Phospholipidic Curcumin: Mirtoselect ® 500 mg tablet, 1000 mg (two oral tablets) per day and Meriva ®, 500 mg tablet, 1000 mg (two oral tablets) per day for 28 days
- Placebo Comparator: placeboA + placeboB per day for four weeks
Period: Overall Study
Arm/Group | Experimental: Anthocyanins+Phospholipidic Curcumin | Placebo Comparator
Started | 17 | 18
Completed | 15 | 14
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Experimental Arm: Mirtoselect ® 500 mg tablet, 1000 mg (two oral tablets) per day, and Meriva ®, 500 mg tablet, 1000 mg (two oral tablets) per day for 28 days
- Control Arm: Placebo A (Mirtoselect® 0 g) + Placebo B (Meriva® 0 gr) /die
- Total: Total of all reporting groups
Arm/Group | Experimental Arm | Control Arm | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (9.8) | 67.9 (10.8) | 69.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 10 | 7 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 14 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Level of Education [Count of Participants; unit: Participants]
  Primary-middle | 5 | 6 | 11
  High university | 10 | 8 | 18
Smoker [Count of Participants; unit: Participants]
  No | 4 | 5 | 9
  Former | 8 | 7 | 15
  Yes | 3 | 2 | 5
Alcholol Habits [Count of Participants; unit: Participants]
  No | 5 | 7 | 12
  Current/Former | 10 | 7 | 17
Baseline BMI [Count of Participants; unit: Participants]
  <25 kg/m^2 | 7 | 9 | 16
  ≥25 kg/m^2 | 8 | 5 | 13
Family history of colorectal cancer [Count of Participants; unit: Participants]
  No | 10 | 7 | 17
  Yes | 5 | 7 | 12
Baseline histological type [Count of Participants; unit: Participants]
  Tubular | 10 | 10 | 20
  Villous | 5 | 4 | 9
Baseline Dysplasia grade [Count of Participants; unit: Participants]
  Low-grade | 12 | 9 | 21
  High-grade | 3 | 5 | 8
# of comorbidity [Median (Inter-Quartile Range); unit: number of comorbidities] | 1 [0 to 3] | 2 [1 to 3] | 2 [1 to 3]
# of concomitant medications [Median (Inter-Quartile Range); unit: number of concomitant medications] | 2 [0 to 4] | 4 [2 to 5] | 3 [1 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Change in Beta Catenin Expression
Description: Change of immunohistochemical expression of beta-catenin in normal and adenomatous colonic tissue
Time Frame: baseline and 4 weeks
Population: Beta-catenin expression according to the treatment arms and the time points in normal tissue and dysplasia
Measure: Mean (Standard Deviation); unit: percentage of positive cells
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 15 | 14
percentage of positive cells
  Pre-treatment: Normal tissue | 100 (0) | 100 (0)
  Pre-treatment: Dysplasia | 100 (0) | 100 (0)
  Post-treatment: Normal tissue | 100 (0) | 100 (0)
  Post-treatment: Dysplasia | 100 (0) | 100 (0)

2. Secondary Outcome: Change in Biomarkes Expression
Description: Change in immunohistochemical expression of Nuclear Factor-Kβ (NFKβ), Ki-67 Labeling Index, and P53 in normal tissue and displasia
Time Frame: baseline and 4 weeks
Population: Tissue biomarker expression according to the treatment arms and the timepoints in normal tissue and dysplasia
Measure: Mean (Standard Deviation); unit: percentage of positive cells
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 15 | 14
percentage of positive cells
  NFKβ Pre-treatment: Normal tissue | 36.7 (21.3) | 52.7 (20.9)
  NFKβ Post-treatment: Normal tissue | 42.3 (31.7) | 50.7 (26.7)
  NFKβ Pre-treatment: Dysplasia | 69.7 (17.2) | 74.3 (15)
  NFKβ Post-treatment: Dysplasia | 74.3 (21.5) | 81.4 (13.5)
  Ki-67 Pre-treatment: Normal tissue | 19.4 (14.6) | 21.2 (11.4)
  Ki-67 Post-treatment: Normal tissue | 16.1 (11.1) | 15.9 (10.5)
  Ki-67 Pre-treatment: Dysplasia | 44.9 (26.4) | 42.9 (19.5)
  Ki-67 Post-treatment: Dysplasia | 58.0 (26.0) | 58.2 (23.6)
  P53 Pre-treatment: Normal tissue | 8.7 (11.4) | 3.5 (4.8)
  P53 Post-treatment: Normal tissue | 3.9 (4.4) | 5.4 (7.3)
  P53 Pre-treatment: Dysplasia | 50.0 (24.2) | 37.5 (20.5)
  P53 Post-treatment: Dysplasia | 60.3 (27.7) | 51.8 (24.1)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Experimental Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 3/15 | 2/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Arm (N=15) | Control Arm (N=14)
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT01948661/Prot_SAP_000.pdf